CLINICAL TRIAL: NCT05117853
Title: The Use of Autofluorescence and Indocyanine Green to Avoid Hypocalcemia After Total Thyroidectomy: A Randomized Clinical Trial
Brief Title: Autofluorescence and Indocyanine Green to Avoid Hypocalcemia After Thyroidectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Responsible Party: Principal Investigator, Klaas Van Den Heede, Principal Investigator / Scientific Fellow, Onze Lieve Vrouw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B1262021000021
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Thyroid Disease; Hypoparathyroidism Postprocedural
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Intervention Model Description: Single-center, comparative, randomized, single-blind, controlled trial against the gold standard of visual identification and viability evaluation.
Who Masked: Participant
Masking Description: Simple blind (Only participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Autofluorescent detection and injection of indocyanine green (Experimental): Drug: indocyanine green (ICG)
  Autofluorescence detection of the parathyroid glands and injection of indocyanine green at two predefined timepoints will be performed to evaluate the vascularization of the parathyroid glands.
  Interventions: Drug: Autofluorescent detection + Injection of indocyanine green
- Control group (Placebo Comparator): Gold standard of visual identification and evaluation of viability.
  Interventions: Procedure: Gold standard of visual identification and evaluation of viability of the parathyroid glands.

INTERVENTIONS:
Drug: Autofluorescent detection + Injection of indocyanine green — All four parathyroid glands will be actively sought for in every case selected for the use of AF/ICG, with AF verification of parathyroid tissue.
  The timepoints of AF will be:
  * 1 = after lateral dissection side 1 (side 1)
  * 2= after lateral dissection side 2 (side 2)
  The timepoints of ICG injection will be:
  * 1 = after the first thyroid lobectomy (side 1)
  * 2 = after the second thyroid lobectomy (side 2)
  Scoring of the viability of parathyroid glands (adapted from Vidal Fortuny et al., 2016):
  * 1 = black = not viable/vascularized
  * 2 = grey = moderately viably/ moderately vascularized
  * 3 = white = viable/well-vascularized
  Other Names: ICG Injection
  Arms: Autofluorescent detection and injection of indocyanine green
Procedure: Gold standard of visual identification and evaluation of viability of the parathyroid glands. — Gold standard of visual identification and evaluation of viability of the parathyroid glands.
  Arms: Control group

SUMMARY:
* Hypoparathyroidism (and the resulting hypocalcemia) remains the most common morbidity after a total thyroidectomy.
* The identification and preservation of parathyroid glands during neck surgery has always been challenging but is crucial to avoid postoperative hypocalcemia.
* Recently, the specific autofluorescent characteristics of endogenous fluorophores in the parathyroid tissue have been used to detect and confirm parathyroid glands during thyroid surgery.
* Injecting indocyanine green and using its fluorescent characteristics has the advantage of adding information about the vascular supply of the parathyroid glands.
* This randomized clinical trial aims to investigate whether using autofluorescence and indocyanine green during thyroid surgery can predict or prevent postoperative hypocalcemia.

DETAILED DESCRIPTION:
Hypoparathyroidism (and the resulting hypocalcemia) remains the most common morbidity after a total thyroidectomy. When defined as corrected serum calcium levels below 2.10 mmol/L, the temporary rates of hypocalcemia after a total thyroidectomy excluding lymph node neck dissection still easily exceed 20% (BAETS fifth national audit report, 2017). When extending the follow-up period to more than six months after surgery, late or permanent hypocalcemia is seen in over 5% of patients after a total thyroidectomy. These British numbers have been confirmed in large European and American databases. A large, Belgian, single-center analysis, including redo-surgery and lymph node neck dissections, confirmed temporary and permanent rates of hypocalcemia of 32% and 3%, respectively.

While temporary hypocalcemia results in a reduced quality of life, additional medical costs to the patients and the society, and hypocalcemia-related symptoms, permanent hypocalcemia adds an increased risk of developing renal failure, basal ganglia calcifications, neuropsychiatric derangements, and infections.

The identification and preservation of parathyroid glands during neck surgery has always been challenging but is crucial to avoid postoperative hypocalcemia. The visual evaluation of parathyroid gland vascularization is even more challenging, prone to subjectivity, and depending on surgical experience and surgical volume. Moreover, even experienced endocrine surgeons appear to be unreliable in using visual scores to assess the viability of parathyroid glands.

Recently, the specific autofluorescent characteristics of endogenous fluorophores in the parathyroid tissue have been used to detect and confirm parathyroid glands during thyroid surgery. However, this signal does not provide any information on viability and vascularization of the parathyroid glands. Injecting indocyanine green (ICG) and using its fluorescent characteristics has the advantage of adding information about the vascular supply of the parathyroid glands. The combined technique of autofluorescent and ICG-enhanced imaging suffers from lack of standardization, optimal technique, dosage, and timing of the ICG administration, and still must prove its possible benefit in a clinical setting.

Hence, this randomized clinical trial aims to investigate whether using autofluorescence (AF) and indocyanine green during thyroid surgery can predict or prevent postoperative hypocalcemia. By using parathyroid gland detection via autofluorescence imaging and verifying their viability after ICG injection, the authors aim to identify patients at risk of hypocalcemia.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients undergoing a total thyroidectomy without previous neck surgery.

Exclusion Criteria:

* Children and teenagers (<18 years old)
* Patients refusing participation or unable/unwilling to sign the informed consent
* Patients with a completion thyroidectomy
* Patients with planned central and lateral neck lymph node dissections (thyroid cancer)
* Patients with previous neck surgery
* Patients with a known allergy/hypersensitivity to indocyanine green

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative hypocalcemia | One week after surgery
  Defined as parathyroid hormone (PTH) levels <15 pg/mL, serum calcium levels <2.10 mmol/L, or the intake of calcium or activated vitamin D supplements after total thyroidectomy.

SECONDARY OUTCOMES:
The number of identified parathyroid glands | 1 hour after surgery
  Visual identification and confirmation with autofluorescence
The number of reimplanted parathyroid glands | 1 hour after surgery
  Visual identification and decision to re-implant after ICG
The presence of late or permanent hypocalcemia | Six months after surgery
  Defined as persistent PTH levels <15 pg/mL, persistent serum calcium levels <2.10 mmol/L, or continued intake of calcium or activated vitamin D supplements more than six months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Onze Lieve Vrouw Hospital, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available from 1 year after till 20 years after final study completion.
Access Criteria: Data access request will be reviewed by the ethics committee of the Onze Lieve Vrouw Hospital, Aalst. Any request will require signing and completing a data access agreement.

REFERENCES:
- [Background] Sitges-Serra A. Etiology and Diagnosis of Permanent Hypoparathyroidism after Total Thyroidectomy. J Clin Med. 2021 Feb 2;10(3):543. doi: 10.3390/jcm10030543. PMID 33540657
- [Background] Moten AS, Thibault DP, Willis AW, Willis AI. Demographics, disparities, and outcomes in substernal goiters in the United States. Am J Surg. 2016 Apr;211(4):703-9. doi: 10.1016/j.amjsurg.2015.11.022. Epub 2016 Jan 6. PMID 26813846
- [Background] Edafe O, Antakia R, Laskar N, Uttley L, Balasubramanian SP. Systematic review and meta-analysis of predictors of post-thyroidectomy hypocalcaemia. Br J Surg. 2014 Mar;101(4):307-20. doi: 10.1002/bjs.9384. Epub 2014 Jan 9. PMID 24402815
- [Background] Lorente-Poch L, Sancho JJ, Munoz-Nova JL, Sanchez-Velazquez P, Sitges-Serra A. Defining the syndromes of parathyroid failure after total thyroidectomy. Gland Surg. 2015 Feb;4(1):82-90. doi: 10.3978/j.issn.2227-684X.2014.12.04. PMID 25713783
- [Background] Van Slycke S, Van Den Heede K, Bruggeman N, Vermeersch H, Brusselaers N. Risk factors for postoperative morbidity after thyroid surgery in a PROSPECTIVE cohort of 1500 patients. Int J Surg. 2021 Apr;88:105922. doi: 10.1016/j.ijsu.2021.105922. Epub 2021 Mar 25. PMID 33774174
- [Background] Van Den Heede K, Tolley NS, Di Marco AN, Palazzo FF. Differentiated Thyroid Cancer: A Health Economic Review. Cancers (Basel). 2021 May 7;13(9):2253. doi: 10.3390/cancers13092253. PMID 34067214
- [Background] Eismontas V, Slepavicius A, Janusonis V, Zeromskas P, Beisa V, Strupas K, Dambrauskas Z, Gulbinas A, Martinkenas A. Predictors of postoperative hypocalcemia occurring after a total thyroidectomy: results of prospective multicenter study. BMC Surg. 2018 Aug 9;18(1):55. doi: 10.1186/s12893-018-0387-2. PMID 30092793
- [Background] Ji YB, Song CM, Sung ES, Jeong JH, Lee CB, Tae K. Postoperative Hypoparathyroidism and the Viability of the Parathyroid Glands During Thyroidectomy. Clin Exp Otorhinolaryngol. 2017 Sep;10(3):265-271. doi: 10.21053/ceo.2016.00724. Epub 2016 Aug 13. PMID 27515510
- [Background] Van Slycke S, Van Den Heede K, Brusselaers N, Vermeersch H. Feasibility of Autofluorescence for Parathyroid Glands During Thyroid Surgery and the Risk of Hypocalcemia: First Results in Belgium and Review of the Literature. Surg Innov. 2021 Aug;28(4):409-418. doi: 10.1177/1553350620980263. Epub 2020 Dec 29. PMID 33372584
- [Background] Benmiloud F, Godiris-Petit G, Gras R, Gillot JC, Turrin N, Penaranda G, Noullet S, Chereau N, Gaudart J, Chiche L, Rebaudet S. Association of Autofluorescence-Based Detection of the Parathyroid Glands During Total Thyroidectomy With Postoperative Hypocalcemia Risk: Results of the PARAFLUO Multicenter Randomized Clinical Trial. JAMA Surg. 2020 Feb 1;155(2):106-112. doi: 10.1001/jamasurg.2019.4613. PMID 31693081
- [Background] Spartalis E, Ntokos G, Georgiou K, Zografos G, Tsourouflis G, Dimitroulis D, Nikiteas NI. Intraoperative Indocyanine Green (ICG) Angiography for the Identification of the Parathyroid Glands: Current Evidence and Future Perspectives. In Vivo. 2020 Jan-Feb;34(1):23-32. doi: 10.21873/invivo.11741. PMID 31882459
- [Background] Riley RD, Moons KGM, Snell KIE, Ensor J, Hooft L, Altman DG, Hayden J, Collins GS, Debray TPA. A guide to systematic review and meta-analysis of prognostic factor studies. BMJ. 2019 Jan 30;364:k4597. doi: 10.1136/bmj.k4597. No abstract available. PMID 30700442
- [Background] Alander JT, Kaartinen I, Laakso A, Patila T, Spillmann T, Tuchin VV, Venermo M, Valisuo P. A review of indocyanine green fluorescent imaging in surgery. Int J Biomed Imaging. 2012;2012:940585. doi: 10.1155/2012/940585. Epub 2012 Apr 22. PMID 22577366
- [Background] Reinhart MB, Huntington CR, Blair LJ, Heniford BT, Augenstein VA. Indocyanine Green: Historical Context, Current Applications, and Future Considerations. Surg Innov. 2016 Apr;23(2):166-75. doi: 10.1177/1553350615604053. Epub 2015 Sep 10. PMID 26359355
- [Background] Obana A, Miki T, Hayashi K, Takeda M, Kawamura A, Mutoh T, Harino S, Fukushima I, Komatsu H, Takaku Y, et al. Survey of complications of indocyanine green angiography in Japan. Am J Ophthalmol. 1994 Dec 15;118(6):749-53. doi: 10.1016/s0002-9394(14)72554-1. PMID 7977601
- [Background] Desmettre T, Devoisselle JM, Mordon S. Fluorescence properties and metabolic features of indocyanine green (ICG) as related to angiography. Surv Ophthalmol. 2000 Jul-Aug;45(1):15-27. doi: 10.1016/s0039-6257(00)00123-5. PMID 10946079
- [Background] Vidal Fortuny J, Belfontali V, Sadowski SM, Karenovics W, Guigard S, Triponez F. Parathyroid gland angiography with indocyanine green fluorescence to predict parathyroid function after thyroid surgery. Br J Surg. 2016 Apr;103(5):537-43. doi: 10.1002/bjs.10101. Epub 2016 Feb 11. PMID 26864909
- [Background] Mirallie E, Borel F, Tresallet C, Hamy A, Mathonnet M, Lifante JC, Brunaud L, Menegaux F, Hardouin JB, Blanchard C; THYRQOL Group; Ansquer C, Mourrain-Langlois E, Delemazure AS, Perrot B, Longhi M, Nomine C, Espitalier F, Drui D, Caillard C, Renaud-Moreau N, Marret O, Mucci S, Christou N. Impact of total thyroidectomy on quality of life at 6 months: the prospective ThyrQoL multicentre trial. Eur J Endocrinol. 2020 Feb;182(2):195-205. doi: 10.1530/EJE-19-0587. PMID 31804967
- [Background] Watt T, Cramon P, Hegedus L, Bjorner JB, Bonnema SJ, Rasmussen AK, Feldt-Rasmussen U, Groenvold M. The thyroid-related quality of life measure ThyPRO has good responsiveness and ability to detect relevant treatment effects. J Clin Endocrinol Metab. 2014 Oct;99(10):3708-17. doi: 10.1210/jc.2014-1322. Epub 2014 Jul 8. PMID 25004246
- [Background] Chen Z, Zhao Q, Du J, Wang Y, Han R, Xu C, Chen X, Shu M. Risk factors for postoperative hypocalcaemia after thyroidectomy: A systematic review and meta-analysis. J Int Med Res. 2021 Mar;49(3):300060521996911. doi: 10.1177/0300060521996911. PMID 33779362
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Tu C, Benn EKT. RRApp, a robust randomization app, for clinical and translational research. J Clin Transl Sci. 2017 Dec;1(6):323-327. doi: 10.1017/cts.2017.310. Epub 2018 Feb 19. PMID 29707253